CLINICAL TRIAL: NCT01999673
Title: SUNRISE: A Phase III, Randomized, Double-Blind, Placebo-Controlled Multicenter Trial of Bavituximab Plus Docetaxel Versus Docetaxel Alone in Patients With Previously Treated Stage IIIb/IV Non-Squamous Non Small-Cell Lung Cancer
Brief Title: Phase 3 Study of Bavituximab Plus Docetaxel Versus Docetaxel Alone in Patients With Late-stage Non-squamous Non-small-cell Lung Cancer
Acronym: SUNRISE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Peregrine Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PPHM 1202; 2013-003953-13 (EudraCT Number)
Record Dates: First submitted 2013-11-25; First posted 2013-12-03 (Estimated); Last update posted 2017-04-21 (Actual); Status verified 2017-04

CONDITIONS: Non-Small-Cell Lung Cancer Stage IIIB; Non-Small-Cell Lung Cancer Stage IV; Non-Small-Cell Lung Cancer Metastatic; Carcinoma, Non-Small-Cell Lung; Non-Small Cell Lung Cancer; Non-Small-Cell Lung Carcinoma; Nonsmall Cell Lung Cancer
Keywords: SUNRISE; PPHM 1202; Bavituximab; Peregrine
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — bavituximab; Docetaxel

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- bavituximab plus docetaxel (Experimental): Six 21-day cycles of docetaxel plus weekly bavituximab. Patients who have not experienced disease progression will continue to receive bavituximab weekly until progression.
  Interventions: Biological: bavituximab; Drug: Docetaxel
- placebo plus docetaxel (Placebo Comparator): Six 21-day cycles of docetaxel plus weekly placebo. Patients who have not experienced disease progression will continue to receive placebo weekly until progression.
  Interventions: Drug: Docetaxel; Other: Placebo (for bavituximab)

INTERVENTIONS:
Biological: bavituximab
  Arms: bavituximab plus docetaxel
Drug: Docetaxel
  Other Names: Taxotere
Other: Placebo (for bavituximab)
  Arms: placebo plus docetaxel

SUMMARY:
The primary purpose of this research study is to see whether adding bavituximab (an investigational drug) to the standard chemotherapy drug docetaxel, will improve the results of the treatment for non-small-cell lung cancer.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female at least 18 years of age
* Histologically or cytologically confirmed and documented stage IIIb/IV non-squamous NSCLC according to the American Joint Committee on Cancer Staging Manual (7th Edition)
* Radiographic disease recurrence or progression during or after front-line platinum-based doublet chemotherapy. For patients with known epidermal growth factor receptor (EGFR) activating mutations or anaplastic lymphoma kinase (ALK) translocations, appropriate targeted treatment should have been used. Mutation testing is not required.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Adequate hematologic, renal and hepatic function

Exclusion Criteria:

* Squamous, small cell, carcinoid, adenosquamous, large-cell neuroendocrine, or mixed histology containing small-cell or squamous-cell NSCLC
* Known history of bleeding disorders, eg, von Willebrand disease or hemophilia
* Cavitary tumors or tumors invading or abutting large blood vessels
* Clinically significant bleeding such as gross hematuria, GI bleeding, and hemoptysis within the 6 months before screening
* Thromboembolic events (eg, deep vein thrombosis, pulmonary embolism, arterial thrombosis) within 6 months of screening
* Grade 2 or higher peripheral neuropathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 582 (Estimated)
Dates: Start 2013-12; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Overall Survival | Approximately up to 36 months

SECONDARY OUTCOMES:
Progression-free survival | Approximately up to 36 months
Overall Response Rate | Approximately up to 36 months
Safety | Approximately up to 36 months
  As measured by adverse event rates and laboratory evaluations

CONTACTS AND LOCATIONS:
Locations (141):
- United States (37):
  - Peregrine Pharmaceuticals Investigational Site, Huntsville, Alabama
  - Peregrine Pharmaceuticals Investigational Site, Chandler, Arizona
  - Peregrine Pharmaceuticals Investigational Site, Glendale, Arizona
  - Peregrine Pharmaceuticals Investigational Site, Greenbrae, California
  - Peregrine Pharmaceuticals Investigational Site, Los Angeles, California
  - Peregrine Pharmaceuticals Investigational Site, Oceanside, California
  - Peregrine Pharmaceuticals Investigational Site, Orange, California
  - Peregrine Pharmaceuticals Investigational Site, West Hills, California
  - Peregrine Pharmaceuticals Investigational Site, Fort Myers, Florida
  - Peregrine Pharmaceuticals Investigational Site, St. Petersburg, Florida
  - Peregrine Pharmaceuticals Investigational Site, Tampa, Florida
  - Peregrine Pharmaceuticals Investigational Site, Athens, Georgia
  - Peregrine Pharmaceuticals Investigational Site, Savannah, Georgia
  - Peregrine Pharmaceuticals Investigational Site, Chicago, Illinois
  - Peregrine Pharmaceuticals Investigational Site, Indianapolis, Indiana
  - Peregrine Pharmaceuticals Investigational Site, Marrero, Louisiana
  - Peregrine Pharmaceuticals Investigational Site, Shreveport, Louisiana
  - Peregrine Pharmaceuticals Investigational Site, Baltimore, Maryland
  - Peregrine Pharmaceuticals Investigational Site, Frederick, Maryland
  - Peregrine Pharmaceuticals Investigational Site, Boston, Massachusetts
  - Peregrine Pharmaceuticals Investigational Site, Lincoln, Nebraska
  - Peregrine Pharmaceuticals Investigational Site, Lebanon, New Hampshire
  - Peregrine Pharmaceuticals Investigational Site, Albuquerque, New Mexico
  - Peregrine Pharmaceuticals Investigational Site, Winston-Salem, North Carolina
  - Peregrine Pharmaceuticals Investigational Site, Cincinnati, Ohio
  - Peregrine Pharmaceuticals Investigational Site, Middletown, Ohio
  - Peregrine Pharmaceuticals Investigational Site, Portland, Oregon
  - Peregrine Pharmaceuticals Investigational Site, Hershey, Pennsylvania
  - Peregrine Pharmaceuticals Investigational Site, Pittsburgh, Pennsylvania
  - Peregrine Pharmaceuticals Investigational Site, Chattanooga, Tennessee
  - Peregrine Pharmaceuticals Investigational Site, Knoxville, Tennessee
  - Peregrine Pharmaceuticals Investigational Site, Nashville, Tennessee
  - Peregrine Pharmaceuticals Investigational Site, Abilene, Texas
  - Peregrine Pharmaceuticals Investigational Site, Dallas, Texas
  - Peregrine Pharmaceuticals Investigational Site, Fort Worth, Texas
  - Peregrine Pharmaceuticals Investigational Site, Temple, Texas
  - Peregrine Pharmaceuticals Investigational Site, Seattle, Washington
- Australia (9):
  - Peregrine Pharmaceuticals Investigational Site, Campbelltown, New South Wales
  - Peregrine Pharmaceuticals Investigational Site, Camperdown, New South Wales
  - Peregrine Pharmaceuticals Investigational Site, Tweed Heads, New South Wales
  - Peregrine Pharmaceuticals Investigational Site, Milton, Queensland
  - Peregrine Pharmaceuticals Investigational Site, Redcliffe, Queensland
  - Peregrine Pharmaceuticals Investigational Site, Elizabeth Vale, South Australia
  - Peregrine Pharmaceuticals Investigational Site, Toorak Gardens, South Australia
  - Peregrine Pharmaceuticals Investigational Site, Geelong, Victoria
  - Peregrine Pharmaceuticals Investigational Site, Wodonga, Victoria
- Belgium (7):
  - Peregrine Pharmaceuticals Investigational Site, Antwerp
  - Peregrine Pharmaceuticals Investigational Site, Brussels
  - Peregrine Pharmaceuticals Investigational Site, Ghent
  - Peregrine Pharmaceuticals Investigational Site, Herstal
  - Peregrine Pharmaceuticals Investigational Site, Liège
  - Peregrine Pharmaceuticals Investigational Site, Mechelen
  - Peregrine Pharmaceuticals Investigational Site, Namur
- France (9):
  - Peregrine Pharmaceuticals Investigational Site, Marseille, Bouches-du-Rhone
  - Peregrine Pharmaceuticals Investigational Site, Caen, Calvados
  - Peregrine Pharmaceuticals Investigational Site, Brest, Finistere
  - Peregrine Pharmaceuticals Investigational Site, Nantes, Loire-Atlantique
  - Peregrine Pharmaceuticals Investigational Site, Nancy, Meurthe-et-Moselle
  - Peregrine Pharmaceuticals Investigational Site, Bayonne, Pyrenees-Atlantiques
  - Peregrine Pharmaceuticals Investigational Site, Rennes
  - Peregrine Pharmaceuticals Investigational Site, Saint-Herblain
  - Peregrine Pharmaceuticals Investigational Site, Saint-Priest-en-Jarez
- Germany (14):
  - Peregrine Pharmaceuticals Investigational Site, Karlsruhe, Baden-Wurttemberg
  - Peregrine Pharmaceuticals Investigational Site, München, Bavaria
  - Peregrine Pharmaceuticals Investigational Site, Immenhausen, Hesse
  - Peregrine Pharmaceuticals Investigational Site, Marburg, Hesse
  - Peregrine Pharmaceuticals Investigational Site, Cologne, North Rhine-Westphalia
  - Peregrine Pharmaceuticals Investigational Site, Erfurt, Thuringia
  - Peregrine Pharmaceuticals Investigational Site, Berlin
  - Peregrine Pharmaceuticals Investigational Site, Großhansdorf
  - Peregrine Pharmaceuticals Investigational Site, Halle
  - Peregrine Pharmaceuticals Investigational Site, Hamburg
  - Peregrine Pharmaceuticals Investigational Site, Kassel
  - Peregrine Pharmaceuticals Investigational Site, Mainz
  - Peregrine Pharmaceuticals Investigational Site, Münster
  - Peregrine Pharmaceuticals Investigational Site, Villingen-Schwenningen
- Greece (9):
  - Peregrine Pharmaceuticals Investigational Site, Pátrai, Achaia
  - Peregrine Pharmaceuticals Investigational Site, Neo Faliro, Athens
  - Peregrine Pharmaceuticals Investigational Site, Athens, Attica
  - Peregrine Pharmaceuticals Investigational Site, Chania, Crete
  - Peregrine Pharmaceuticals Investigational Site, Heraklion, Irakleio
  - Peregrine Pharmaceuticals Investigational Site, Thermi, Thessaloniki
  - Peregrine Pharmaceuticals Investigational Site, Athens
  - Peregrine Pharmaceuticals Investigational Site, Larissa
  - Peregrine Pharmaceuticals Investigational Site, Thessaloniki
- Hungary (6):
  - Peregrine Pharmaceuticals Investigational Site, Budapest
  - Peregrine Pharmaceuticals Investigational Site, Győr
  - Peregrine Pharmaceuticals Investigational Site, Gyula
  - Peregrine Pharmaceuticals Investigational Site, Szolnok
  - Peregrine Pharmaceuticals Investigational Site, Törökbálint
  - Peregrine Pharmaceuticals Investigational Site, Zalaegerszeg
- Italy (10):
  - Peregrine Pharmaceuticals Investigational Site, Meldola, Forli-Cesena
  - Peregrine Pharmaceuticals Investigational Site, Lido di Camaiore, Lucca
  - Peregrine Pharmaceuticals Investigational Site, Taormina, Messina
  - Peregrine Pharmaceuticals Investigational Site, Monza, Monza Brianza
  - Peregrine Pharmaceuticals Investigational Site, Aviano, Pordenone
  - Peregrine Pharmaceuticals Investigational Site, Bergamo
  - Peregrine Pharmaceuticals Investigational Site, Cremona
  - Peregrine Pharmaceuticals Investigational Site, Genova
  - Peregrine Pharmaceuticals Investigational Site, Milan
  - Peregrine Pharmaceuticals Investigational Site, Turin
- Romania (5):
  - Peregrine Pharmaceuticals Investigational Site, Brasov
  - Peregrine Pharmaceuticals Investigational Site, Cluj-Napoca
  - Peregrine Pharmaceuticals Investigational Site, Ploieşti
  - Peregrine Pharmaceuticals Investigational Site, Suceava
  - Peregrine Pharmaceuticals Investigational Site, Turda
- Russia (6):
  - Peregrine Pharmaceuticals Investigational Site, Kursk
  - Peregrine Pharmaceuticals Investigational Site, Nizhny Novgorod
  - Peregrine Pharmaceuticals Investigational Site, Obninsk
  - Peregrine Pharmaceuticals Investigational Site, Saint Petersburg
  - Peregrine Pharmaceuticals Investigational Site, Yaroslavl
  - Peregrine Pharmaceuticals Investigational Site, Yekaterinburg
- South Korea (7):
  - Peregrine Pharmaceuticals Investigational Site, Suwon, Gyeonggi-do
  - Peregrine Pharmaceuticals Investigational Site, Suwon, Gyonggi-do
  - Peregrine Pharmaceuticals Investigational Site, Busan
  - Peregrine Pharmaceuticals Investigational Site, Cheongju-si
  - Peregrine Pharmaceuticals Investigational Site, Incheon
  - Peregrine Pharmaceuticals Investigational Site, Seongnam
  - Peregrine Pharmaceuticals Investigational Site, Seoul
- Spain (10):
  - Peregrine Pharmaceuticals Investigational Site, Badalona, Barcelona
  - Peregrine Pharmaceuticals Investigational Site, L'Hospitalet de Llobregat, Barcelona
  - Peregrine Pharmaceuticals Investigational Site, Manresa, Barcelona
  - Peregrine Pharmaceuticals Investigational Site, Majadahonda, Madrid
  - Peregrine Pharmaceuticals Investigational Site, Pamplona, Navarre
  - Peregrine Pharmaceuticals Investigational Site, A Coruña
  - Peregrine Pharmaceuticals Investigational Site, Barcelona
  - Peregrine Pharmaceuticals Investigational Site, Madrid
  - Peregrine Pharmaceuticals Investigational Site, Málaga
  - Peregrine Pharmaceuticals Investigational Site, Valencia
- Taiwan (6):
  - Peregrine Pharmaceuticals Investigational Site, Kaohsiung City
  - Peregrine Pharmaceuticals Investigational Site, Putzu
  - Peregrine Pharmaceuticals Investigational Site, Taichung
  - Peregrine Pharmaceuticals Investigational Site, Tainan
  - Peregrine Pharmaceuticals Investigational Site, Taipei
  - Peregrine Pharmaceuticals Investigational Site, Taoyuan District
- Ukraine (6):
  - Peregrine Pharmaceuticals Investigational Site, Chernivtsi
  - Peregrine Pharmaceuticals Investigational Site, Dnipropetrovsk
  - Peregrine Pharmaceuticals Investigational Site, Khmelnytskyi
  - Peregrine Pharmaceuticals Investigational Site, Kyiv
  - Peregrine Pharmaceuticals Investigational Site, Lutsk
  - Peregrine Pharmaceuticals Investigational Site, Uzhhorod

REFERENCES:
- [Derived] Gerber DE, Horn L, Boyer M, Sanborn R, Natale R, Palmero R, Bidoli P, Bondarenko I, Germonpre P, Ghizdavescu D, Kotsakis A, Lena H, Losonczy G, Park K, Su WC, Tang M, Lai J, Kallinteris NL, Shan JS, Reck M, Spigel DR. Randomized phase III study of docetaxel plus bavituximab in previously treated advanced non-squamous non-small-cell lung cancer. Ann Oncol. 2018 Jul 1;29(7):1548-1553. doi: 10.1093/annonc/mdy177. PMID 29767677